CLINICAL TRIAL: NCT00495846
Title: Treatment of Advanced Hepatocellular Carcinoma With Depot Somatostatin Analogues: a Pilot Prospective Study Based on Somatostatin Receptors Tumors Expression
Brief Title: GH, IGF-I and Somatostatin Analogues in Hepatocellular Carcinoma
Acronym: SS-HCC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Ospedali dei Colli (Other)
Responsible Party: Annamaria Colao, Federico II U
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-4
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Somatostatin analogues; Somatostatin receptors; Octreotide; Lanreotide; IGF-I; IGF-II
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 1. Patients with cirrhosis without HCC in all liver function classes already receiving specific therapy for cirrhosis who accept be subjected to liver biopsy and to sign the written informed consent to participate to the study
  2. Patients with cirrhosis with multifocal HCC and clinical and/or radiological signs of persistence or recurrence of HCC in presence or absence of trombosis of the portal vein, with a single nodule of >6 cm in size or multiple nodules of >3 cm in size who accept be subjected to liver biopsy and to sign the written informed consent to participate to the study
  Interventions: Drug: Octreotide-LAR, Lanreotide Autogel
- B (Other): Historical controls
  Interventions: Other: Locoregional treatments

INTERVENTIONS:
Drug: Octreotide-LAR, Lanreotide Autogel — Octreotide-LAR intramuscular, dose of 30 mg every 28 days to increase up to 60 mg; lanreotide autogel 120 mg deep subcutaneous every 28 days for 3 months then uptitrated according with the protocol.
  Other Names: Sandostatin-LAR; Ipstyl 120 mg; Somatuline Depot
  Arms: A
Other: Locoregional treatments
  Arms: B

SUMMARY:
The hepatocellular carcinoma (HCC) represents more than 5% of all human malignancies, with more than 500,000 deaths per year (1). In Campania region, mortality for HCC is 2 times higher than in the rest of Italy because of a higher locally prevalence of hepatitis-C virus infection.

Development of HCC in liver cirrhosis is associated with increased DNA synthesis and regeneration of hepatocytes (2). Hepatocyte growth factor, the transforming growth factor-α, the fibroblast growth factor are well studied (3,4) while the insulin-like growth factor system (IGF-I, IGF-II and their binding proteins) has been less investigated. IGF-I and IGF-II modulate growth, metabolism and cell differentiation and have specific receptors in the liver (5). IGF-I levels in the upper normal range have been associated with an increased risk to develop prostate cancer (6), breast cancer (7) and colon cancer (8). Some data report increased expression of IGF-II in HCC (9,10) and others suggest a role of increased IGF-I bioavailability in HCC (11). We reported increased IGF-I/IGFBP-3 ratio in patients with HCC compared with those with cirrhosis with a similar liver function, so suggesting increased IGF-I bioavailability in HCC (12).

There is no currently medical treatment for patients with advanced HCC which has a very poor prognosis (survival <6 months). Because of limited liver function, classical chemotherapy cannot be applied (13). In patients with HCC without cirrhosis, surgery is possible only in 5% while in those with cirrhosis first-line treatment is still questioned as survival is <50% three years after operation. Patients suitable for local resection of HCC are only those with Child-Pugh's "hyper A" liver function class, who are a minority (14-16). Percutaneous resection treatments may treat approximately 70%-90% of tumors with maximal diameters of <3 cm (15,17-19).

Somatostatin analogues are indicated in patients with neuroendocrine tumors expressing somatostatin receptors type 2 and 5 and has excellent safety profile. In advanced HCC, some studies demonstrated beneficial effects (20,21) while some others did not (22,23).

Only a few data are available on somatostatin receptor expression in HCC (24,25). Somatostatin analogues have also a clear-cut inhibitory effect on circulating IGF-I levels with a potential additional effect in delaying HCC progression.

DETAILED DESCRIPTION:
Study objectives

1. To evaluate relationships between GH/IGF-I and IGF-II axis and development and progression of HCC;
2. To evaluate the expression of somatostatin receptor expression in biopsies of HCC by quantitative RT-PCR and immunohistochemistry and in vivo by octreoscan;
3. To evaluate the efficacy of octreotide-LAR or lanreotide-autogel as compared to placebo on clinical symptoms, liver function, biological markers and tumor dimensions by ultrasonography in advanced HCC patients;
4. To correlate the response to somatostatin analogues to somatostatin receptor expression in vitro and in vivo and suppression of the IGF-I and -II axis.

Study design

This is a pilot, open, prospective, monocentric study addressed to:

1. patients with liver cirrhosis and multifocal HCC with or without portal vein invasion;
2. patients with liver cirrhosis and single HCC nodule of >6 cm in size with or without portal vein invasion [principal branch, right branch (one or more segmentary arms), left branch (one or more segmentary arms)];
3. patients with liver cirrhosis and more than 3 HCC nodules of > 3 cm in size with or without portal vein invasion [principal branch, right branch (one or more segmentary arms), left branch (one or more segmentary arms)];
4. patients with cirrhosis without HCC.

Study protocol All enrolled subjects will be subjects to a baseline evaluation and a post-treatment evaluation according with the treatment protocol (see below).

A) Clinical study in vivo diagnostic routine analysis (clinical evaluation, ECG, chest X-ray, blood chemistry, analysis of liver function, α-FP assay, CEA, liver ultrasonography and angio-ultrasonography, abdominal CT scan or MRI); blood sampling for GH, IGF-I, IGF-II, IGFBP-3, ALS, insulin, IGFBP-1 and IGFBP-2; whole body scintigraphy with radiolabeled octreotide (octreoscan) liver biopsy in patients in good clinical condition according with good clinical practice procedures. Biopsy will be performed under ultrasonography guidance with a 19G or 21G needle after local subcutaneous anesthesia (lidocaine 2%). Abdominal ultrasonography will followed biopsy to exclude hemorrage. The tissue sample will be stores at -80° until analysis.

B) Morphological in vitro study the expression of somatostatin receptors will be performed by immunohistochemistry in sequential sections as well as by RT-PCR using specific primers for all receptors; the study includes an analysis of classical histology and immunohistochemical markers. The study includes positive and negative controls for an appropriate analysis of the results.

Study duration

The first study is a pilot study which expected number of patients fulfilling the inclusion criteria is 15 to address the issue of liver cirrhosis with HCC. The enrollment period will be of 12 months or shorter if the 15 patients are enrolled in a shorter time. The observational period is expected to be 3-12 months, according with previous studies. Treatment will be continued in all survivors even if the study will end after 12 months, according with previous studies. Subsequently, the study will proceed with a placebo-controlled randomized study according with the results obtained in the pilot study and will enroll 30-60 in case of patients with HCC without cirrhosis and 20-40 for patients with liver cirrhosis and HCC. All patients will be registered in dedicated CRF and data will be collected by investigators not involved in data analysis.

Withdrawal from the study

The causes of early study withdrawal will be recorded according with:

1. adverse events;
2. no treatment response or patients' clinical condition deterioration according with the investigator judgment;
3. major protocol violation;
4. patient's withdrawal of the consent.

Concomitant therapies All patients will continue all treatments as per investigator judgment. In case some therapy will be withdrawn this will be recorded in the CRF and analyzed as a potential beneficial effect of somatostatin analogues therapy.

Main outcome measures A) Efficacy parameters

For cirrhosis:

Stabilization or improvement of live function parameters Reduction of biological markers of disease (if elevated before starting the treatment) Improvement of quality of life according with SF36 questionnaire

For HCC:

Prolongation of the survival curve (>6 months) Stabilization or reduction of tumor size Reduction or disappearance of portal vein thrombosis Stabilization or improvement of live function parameters Reduction of biological markers of disease (if elevated before starting the treatment) Improvement of quality of life according with SF36 questionnaire

Expected results

The expected results are:

1. Both cirrhotic and normal liver express somatostatin receptors. The different receptor pattern can suggest a role of this receptor subtype in HCC development. The correlation study can also give insight into any role of somatostatin receptors in differentiation, staging and prognosis of HCC.
2. Treatment with somatostatin analogues will prolong survival in advanced HCC patients. This should occur according with liver function before starting the treatment. We expect that patients having tumors with high expression of SS-2 receptors on their HCC will have the longest survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis without HCC in all liver function classes already receiving specific therapy for cirrhosis who accept be subjected to liver biopsy and to sign the written informed consent to participate to the study
* Patients with cirrhosis with multifocal HCC and clinical and/or radiological signs of persistence or recurrence of HCC in presence or absence of thrombosis of the portal vein, with a single nodule of > 6 cm in size or multiple nodules of > 3 cm in size who accept be subjected to liver biopsy and to sign the written informed consent to participate to the study

Exclusion Criteria:

* Age < 18 yrs or > 75 yrs
* Pregnancy or lactation
* Intolerance to somatostatin analogues

Treatment protocol:

* In all patients fulfilling the inclusion criteria, treatment will begin with octreotide-LAR at a dose of 30 mg every 28 days or lanreotide autogel 120 mg every 28 days for 3 months.
* After 28, 56 and 74 days (immediately before the next injection) all patients will be admitted to the Day Hospital of the IX Division of Internal Medicine of the D. Cotugno Hospital for the clinical examination, blood chemistry, blood sampling for the IGF axis analysis, and abdominal ultrasound. After 74 days, abdominal CT or MRI will also be performed.
* Then, in all survivors the interval between injection will be reduced to 21 days and follow up for the next 3 months will be done as stated before the day immediately preceding the injection.
* Then, in the subsequent follow-up the interval between injection will be reduced to 14 days and all procedures will be repeated at monthly intervals.
* All the patients fulfilling the inclusion criteria but refusing to participate to the study will be followed with the same methodology of those receiving the somatostatin analogues treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prolongation of the survival curve (>6 months) | 12 months

SECONDARY OUTCOMES:
Improvement of liver function, Reduction of biological markers of disease (if elevated before starting the treatment) | 12 months
Improvement of quality of life according with SF36 questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, PhD, Principal Investigator — University Federico II of Naples
Locations (1):
- D. Cotugno Hospital, Naples, Italy

REFERENCES:
- [Result] Llovet JM, Beaugrand M. Hepatocellular carcinoma: present status and future prospects. J Hepatol. 2003;38 Suppl 1:S136-49. doi: 10.1016/s0168-8278(02)00432-4. No abstract available. PMID 12591191
- [Result] Blanc P, Desprez D, Fabre JM, Pageaux G, Daures JP, Larrey D, Saint-Aubert B, Michel H, Maurel P. Contribution of primary cultures of adult human hepatocytes to the pathophysiology of hepatocellular carcinoma. J Hepatol. 1996 Nov;25(5):663-9. doi: 10.1016/s0168-8278(96)80236-4. PMID 8938543
- [Result] Burr AW, Hillan KJ, McLaughlin KE, Ferrier R, Chapman C, Mathew J, Burt AD. Hepatocyte growth factor levels in liver and serum increase during chemical hepatocarcinogenesis. Hepatology. 1996 Nov;24(5):1282-7. doi: 10.1002/hep.510240549. PMID 8903411
- [Result] Tomiya T, Fujiwara K. Serum transforming growth factor alpha level as a marker of hepatocellular carcinoma complicating cirrhosis. Cancer. 1996 Mar 15;77(6):1056-60. doi: 10.1002/(sici)1097-0142(19960315)77:63.0.co;2-f. PMID 8635123
- [Result] Jones JI, Clemmons DR. Insulin-like growth factors and their binding proteins: biological actions. Endocr Rev. 1995 Feb;16(1):3-34. doi: 10.1210/edrv-16-1-3. No abstract available. PMID 7758431
- [Result] Chan JM, Stampfer MJ, Giovannucci E, Gann PH, Ma J, Wilkinson P, Hennekens CH, Pollak M. Plasma insulin-like growth factor-I and prostate cancer risk: a prospective study. Science. 1998 Jan 23;279(5350):563-6. doi: 10.1126/science.279.5350.563. PMID 9438850
- [Result] Hankinson SE, Willett WC, Colditz GA, Hunter DJ, Michaud DS, Deroo B, Rosner B, Speizer FE, Pollak M. Circulating concentrations of insulin-like growth factor-I and risk of breast cancer. Lancet. 1998 May 9;351(9113):1393-6. doi: 10.1016/S0140-6736(97)10384-1. PMID 9593409
- [Result] Giovannucci E, Pollak M, Platz EA, Willett WC, Stampfer MJ, Majeed N, Colditz GA, Speizer FE, Hankinson SE. Insulin-like growth factor I (IGF-I), IGF-binding protein-3 and the risk of colorectal adenoma and cancer in the Nurses' Health Study. Growth Horm IGF Res. 2000 Apr;10 Suppl A:S30-1. doi: 10.1016/s1096-6374(00)90014-5. No abstract available. PMID 10984283
- [Result] Nardone G, Romano M, Calabro A, Pedone PV, de Sio I, Persico M, Budillon G, Bruni CB, Riccio A, Zarrilli R. Activation of fetal promoters of insulinlike growth factors II gene in hepatitis C virus-related chronic hepatitis, cirrhosis, and hepatocellular carcinoma. Hepatology. 1996 Jun;23(6):1304-12. doi: 10.1002/hep.510230602. PMID 8675143
- [Result] Yang D, Faris R, Hixson D, Affigne S, Rogler CE. Insulin-like growth factor II blocks apoptosis of N-myc2-expressing woodchuck liver epithelial cells. J Virol. 1996 Sep;70(9):6260-8. doi: 10.1128/JVI.70.9.6260-6268.1996. PMID 8709253
- [Result] Buzzelli G, Dattolo P, Pinzani M, Brocchi A, Romano S, Gentilini P. Circulating growth hormone and insulin-like growth factor-I in nonalcoholic liver cirrhosis with or without superimposed hepatocarcinoma: evidence of an altered circadian rhythm. Am J Gastroenterol. 1993 Oct;88(10):1744-8. PMID 8213718
- [Result] Mattera D, Capuano G, Colao A, Pivonello R, Manguso F, Puzziello A, D'Agostino L. Increased IGF-I : IGFBP-3 ratio in patients with hepatocellular carcinoma. Clin Endocrinol (Oxf). 2003 Dec;59(6):699-706. doi: 10.1046/j.1365-2265.2003.01909.x. PMID 14974910
- [Result] Llovet JM, Fuster J, Bruix J. Intention-to-treat analysis of surgical treatment for early hepatocellular carcinoma: resection versus transplantation. Hepatology. 1999 Dec;30(6):1434-40. doi: 10.1002/hep.510300629. PMID 10573522
- [Result] Llovet JM, Fuster J, Bruix J; Barcelona-Clinic Liver Cancer Group. The Barcelona approach: diagnosis, staging, and treatment of hepatocellular carcinoma. Liver Transpl. 2004 Feb;10(2 Suppl 1):S115-20. doi: 10.1002/lt.20034. PMID 14762851
- [Result] Livraghi T, Goldberg SN, Lazzaroni S, Meloni F, Solbiati L, Gazelle GS. Small hepatocellular carcinoma: treatment with radio-frequency ablation versus ethanol injection. Radiology. 1999 Mar;210(3):655-61. doi: 10.1148/radiology.210.3.r99fe40655. PMID 10207464
- [Result] Livraghi T, Giorgio A, Marin G, Salmi A, de Sio I, Bolondi L, Pompili M, Brunello F, Lazzaroni S, Torzilli G, et al. Hepatocellular carcinoma and cirrhosis in 746 patients: long-term results of percutaneous ethanol injection. Radiology. 1995 Oct;197(1):101-8. doi: 10.1148/radiology.197.1.7568806.
- [Result] Lencioni RA, Allgaier HP, Cioni D, Olschewski M, Deibert P, Crocetti L, Frings H, Laubenberger J, Zuber I, Blum HE, Bartolozzi C. Small hepatocellular carcinoma in cirrhosis: randomized comparison of radio-frequency thermal ablation versus percutaneous ethanol injection. Radiology. 2003 Jul;228(1):235-40. doi: 10.1148/radiol.2281020718. Epub 2003 May 20. PMID 12759473
- [Result] Kouroumalis E, Samonakis D, Skordilis P. Octreotide treatment of hepatocellular carcinoma. Hepatology. 2003 Feb;37(2):477. doi: 10.1053/jhep.2003.50026. No abstract available. PMID 12540801
- [Result] Samonakis DN, Moschandreas J, Arnaoutis T, Skordilis P, Leontidis C, Vafiades I, Kouroumalis E. Treatment of hepatocellular carcinoma with long acting somatostatin analogues. Oncol Rep. 2002 Jul-Aug;9(4):903-7. PMID 12066229
- [Result] Kapadia CR. Somatostatin and hepatocellular carcinoma. Gastroenterology. 1998 Nov;115(5):1298-9. doi: 10.1016/s0016-5085(98)70109-x. No abstract available. PMID 9797392
- [Result] Raderer M, Hejna MH, Muller C, Kornek GV, Kurtaran A, Virgolini I, Fiebieger W, Hamilton G, Scheithauer W. Treatment of hepatocellular cancer with the long acting somatostatin analog lanreotide in vitro and in vivo. Int J Oncol. 2000 Jun;16(6):1197-201. doi: 10.3892/ijo.16.6.1197. PMID 10811995
- [Result] Raderer M, Hejna MH, Kurtaran A, Kornek GV, Valencak JB, Oberhuber G, Vorbeck F, Virgolini I, Scheithauer W. Successful treatment of an advanced hepatocellular carcinoma with the long-acting somatostatin analog lanreotide. Am J Gastroenterol. 1999 Jan;94(1):278-9. doi: 10.1111/j.1572-0241.1999.00821.x. PMID 9934776
- [Result] Yuen MF, Poon RT, Lai CL, Fan ST, Lo CM, Wong KW, Wong WM, Wong BC. A randomized placebo-controlled study of long-acting octreotide for the treatment of advanced hepatocellular carcinoma. Hepatology. 2002 Sep;36(3):687-91. doi: 10.1053/jhep.2002.35071. PMID 12198662
- [Result] Reubi JC, Zimmermann A, Jonas S, Waser B, Neuhaus P, Laderach U, Wiedenmann B. Regulatory peptide receptors in human hepatocellular carcinomas. Gut. 1999 Nov;45(5):766-74. doi: 10.1136/gut.45.5.766. PMID 10517918
- [Result] Blaker M, Schmitz M, Gocht A, Burghardt S, Schulz M, Broring DC, Pace A, Greten H, De Weerth A. Differential expression of somatostatin receptor subtypes in hepatocellular carcinomas. J Hepatol. 2004 Jul;41(1):112-8. doi: 10.1016/j.jhep.2004.03.018. PMID 15246216
- [Result] Dimitroulopoulos D, Xinopoulos D, Tsamakidis K, Zisimopoulos A, Andriotis E, Panagiotakos D, Fotopoulou A, Chrysohoou C, Bazinis A, Daskalopoulou D, Paraskevas E. Long acting octreotide in the treatment of advanced hepatocellular cancer and overexpression of somatostatin receptors: randomized placebo-controlled trial. World J Gastroenterol. 2007 Jun 21;13(23):3164-70. doi: 10.3748/wjg.v13.i23.3164. PMID 17589893
- [Result] Cebon J, Findlay M, Hargreaves C, Stockler M, Thompson P, Boyer M, Roberts S, Poon A, Scott AM, Kalff V, Garas G, Dowling A, Crawford D, Ring J, Basser R, Strickland A, Macdonald G, Green M, Nowak A, Dickman B, Dhillon H, Gebski V; Australasian Gastro-Intestinal Trials Group (AGITG) Ag0001H Investigators. Somatostatin receptor expression, tumour response, and quality of life in patients with advanced hepatocellular carcinoma treated with long-acting octreotide. Br J Cancer. 2006 Oct 9;95(7):853-61. doi: 10.1038/sj.bjc.6603325. Epub 2006 Sep 5. PMID 16953241